CLINICAL TRIAL: NCT05361161
Title: Transarterial Chemoembolization With Lipiodol in the Treatment of Initial Unresectable Gastric Cancer (GC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gang Wu (Other)
Responsible Party: Sponsor-Investigator, Gang Wu, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACE-GC-001
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Gastric Cancer; Embolization
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transarterial Chemoembolization With Lipiodol for Initial Unresectable Gastric Cancer (Experimental)
  Interventions: Drug: Transarterial Chemoembolization

INTERVENTIONS:
Drug: Transarterial Chemoembolization — Arterial infusion chemotherapy (THP + oxaliplatin + raltitrexed) and THP combined with lipiodol embolization for 2 times, with an interval of 1 month.

SUMMARY:
This is a prospective, open-labelled study to evaluate the efficacy and safety of sequential transarterial chemoembolization with lipiodol and neoadjuvant chemotherapy in the treatment of Initial unresectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and imaging diagnosis of gastric adenocarcinoma with initial unresectable R0;
2. Age (18-80 years old) and gender are not limited;
3. No extragastric organ transfer;
4. No serious diseases of the heart, liver, lung, kidney and other organs;
5. Expected survival time > 3 months;
6. Physical performance status score ECOG ≤1 point;
7. Females of reproductive age must have a negative pregnancy test; or male and female patients must agree to use effective contraception during treatment and within 1 year thereafter.

Exclusion Criteria:

1. Poor coagulation function, INR>1.5, or ongoing anticoagulation therapy or known bleeding diseases;
2. WBC <3000/mm3 or platelet count <50000/mm3;
3. AST and/or ALT > 3 times the upper limit of normal;
4. Comorbidities or social environment that can cause subjects to fail to follow the research plan or even endanger patient safety;
5. The patient has other primary tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluation | up to 3 years
  Objective response rate (ORR): complete response (CR) + partial response (PR). Evaluation methods: Objective tumor response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Subjects must have measurable tumor lesions at baseline, and the efficacy evaluation criteria are divided into complete remission (CR), partial remission (PR), stable disease (SD), and progressive disease (PD) according to RECIST 1.1 criteria. Complete Remission (CR): All target and non-target lesions disappeared, no new lesions; Partial Remission (PR): Compared with baseline, tumor burden decreased by ≥30%, and non-target lesions did not progress significantly , no new lesions; Stable Disease (SD): neither PR nor PD; Progressive Disease (PD): tumor burden increased by ≥20%, and the absolute value increased by at least 5mm, or non-target lesions progressed, or new lesions (reconfirm progression after at least 6 weeks).
Surgical resection rate | up to 3 years
  Surgical resection rate: The rate of surgical resection is transformed from those who cannot undergo radical surgical resection and one-stage anastomosis after treatment.
PFS | up to 3 years
  Progression-free survival（PFS） is defined as the time between the date of randomization and any documented tumor progression or death from any cause.
OS | up to 3 years
  Overall survival (OS), defined as the time from study entry (ie, signing the ICF) to death from any cause. For subjects who were alive at the last contact, their overall survival was censored on the date of the last contact.

IPD SHARING:
Plan to Share IPD: No